CLINICAL TRIAL: NCT06697821
Title: The Number of Mesogastria Containing Metastatic Lymph Nodes Predicts Gastric Cancer Prognosis
Status: Completed | Type: Observational
Sponsor: Jichao Qin (Other)
Responsible Party: Sponsor-Investigator, Jichao Qin, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: TJ-IRB202403050
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Gastric Cancer
Keywords: metastasis; Gastric Cancer; Lymph node; Mesogastrium
MeSH Terms: conditions — Stomach Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: D2＋CME — Whether to perform the whole mesogastric excision

SUMMARY:
To investigate the impact of the number of mesogastria containing metastatic lymph nodes on the prognosis of gastric cancer.

DETAILED DESCRIPTION:
Previous studies have established the existence of the mesogastrium, dividing it into six sections. The mesogastrium is identified during surgery and utilized in surgical practice. The aim of the present study was to further investigate its role in gastric cancer prognosis.Between January 2014 and January 2018, patients from the Tongji Hospital were included in this post-hoc analysis, including data from a randomized clinical study (DCGC01; http://www.clinicaltrials.gov, NCT01978444). Mesogastria containing metastatic lymph nodes (LNs) were referred to as metastatic mesogastria. Pathology reports were examined to assess metastases in the mesogastrium. Survival was assessed using Kaplan-Meier curves and multivariable Cox models.

ELIGIBILITY:
Inclusion Criteria:

1. older than 18, younger than 85
2. primary gastric adenocarcinoma confirmed by preoperative pathology
3. routine blood tests, liver and kidney functions and who health status score are within the range of tolerable surgery
4. it is expected to perform radical gastrectomy through d2+cme

Exclusion Criteria:

1. pregnant or lactating women
2. severe mental disorder or language communication disorder
3. preoperative imaging examination or intraoperative exploration found that the patient had the following conditions: tumor involving surrounding organs requiring combined organ resection, distant organ metastasis or R0 resection could not be achieved
4. those who are not suitable for laparoscopic surgery (such as extensive adhesion caused by anterior abdominal surgery and pneumoperitoneum for various reasons).
5. concurrent malignancies at other sites
6. emergency surgery patients

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with gastric cancer who underwent total or proximal gastrectomy in Tongji Hospital were included in this study
Sampling Method: Non-Probability Sample
Enrollment: 480 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | Postoperative 5-year survival
  Postoperative 5-year survival

SECONDARY OUTCOMES:
The Number of Mesogastria Containing Metastatic Lymph Nodes | Postoperative 5-year
  The Number of Mesogastria Containing Metastatic Lymph Nodes

CONTACTS AND LOCATIONS:
Overall Officials: Jichao Qin, M.D./Ph.D, Principal Investigator — Huazhong University of Science and Technology
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No